CLINICAL TRIAL: NCT04684901
Title: A Randomized, Controlled Study to Evaluate Effectiveness of AlloWrap® Amniotic Membrane for the Reduction of Post-Operative Soft Tissue Inflammation in Two-Level Anterior Cervical Discectomy and Fusion Procedures
Brief Title: Effectiveness of AlloWrap® for the Reduction of Inflammation in ACDF Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWR-001
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cervical Stenosis; Spondylolisthesis; Cervical Radiculopathy; Cervical Disc Disorder
Keywords: Anterior Cervical Discectomy and Fusion Surgery; ACDF Surgery
MeSH Terms: conditions — Spondylolisthesis; Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention): Standard of Care - No AlloWrap used during surgery
- AlloWrap Group (Experimental): AlloWrap used in surgery
  Interventions: Other: AlloWrap® Amniotic Membrane

INTERVENTIONS:
Other: AlloWrap® Amniotic Membrane — AlloWrap is a human amniotic membrane designed to provide a biologic barrier following surgical repair.
  Arms: AlloWrap Group

SUMMARY:
The primary objective of this study is to obtain evidence of the effectiveness of AlloWrap Amniotic Membrane in the reduction of soft tissue swelling in two-level ACDF procedures.

DETAILED DESCRIPTION:
AlloWrap® is a dual sided human amniotic membrane, procured from consented human tissue donors who elect to have scheduled cesarean births. A Human Cells, Tissues, and Cellular and Tissue-Based Product (HCT/P) as defined by the United States Food and Drug Administration (FDA) 21 CFR Part 1271, AlloWrap® is intended to provide a biologic barrier following surgical repair. Designed to meet the clinical needs of the patient and practical needs of the clinical setting amniotic based surgical barriers have been shown to contain a natural balance of cytokines that can assist the body in reducing epidural fibrosis, inflammation, and infection at the surgical site. Using AlloWrap® as a surgical barrier may result in outcomes with less scaring, potentially reducing pain and assisting the patient in returning to normal functionality while potentially making revision dissections less complicated. The purpose of this clinical study is to evaluate the use of AlloWrap® Amniotic Membrane in ACDF procedures to obtain evidence of effectiveness, defined as the reduction, and the possible prevention, of complications associated with ACDF surgery such as odynophagia and/or dysphasia that result from soft tissue inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Be a skeletally mature male or a non-pregnant, non-lactating female ≥18 years of age;
* Radiographically diagnosed with cervical stenosis or cervical disc disorder and/or degeneration, spondylolisthesis and/or cervical radiculopathy resulting from neural element compression as confirmed by MRI, CT, CT myelogram;
* Neurological dysfunction or radicular symptoms by history and physical exam;
* Is scheduled/or will be scheduled to undergo an anterior cervical fusion, requiring internal fixation using an anterior cervical standalone interbody cage system;
* Failed to gain adequate relief from non-operative treatment, including but not limited to medications, physical therapy, chiropractic care, home exercise and/or for at least 6 weeks; or the patient has progressive muscle weakness or atrophy or intractable pain;
* Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.

Exclusion Criteria:

* Have a documented medical history or radiographic evidence of osteoporosis or other condition which would negatively impact the bone healing process (e.g. history of Paget's disease, osteomalacia, or other osteodystrophy) or preclude the subject from receiving screw fixation;
* Have had or plans to have an epidural steroid injection or has taken NSAIDs ≤ 7 days prior to surgery;
* Circulatory, cardiac, or pulmonary problems that could cause excessive surgical risk based on the opinion of the Investigator;
* Active malignancy; Nondiscogenic source of symptoms (e.g., tumor, etc.) or undergoing treatment for tumor or boney traumatic injury to the cervical spine or a history of any invasive malignancy (except non-melanoma skin cancer), unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
* Acute cervical trauma ≤ 6 months prior to surgery;
* Inflammatory disease of the cervical spine;
* Has a history of substance abuse (recreational drugs, alcohol) that has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an in-patient substance abuse program;
* Is currently involved in a study of another investigational product for similar purpose or has been in the previous 90 days;
* Active infection at the operative level, or a systemic infection including prior or pending treatment for HIV, Hepatitis B or Hepatitis C;
* Mentally compromised (e.g., being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease) in a manner that would compromise his or her ability to participate in the clinical study;
* Currently immunologically suppressed or immunocompromised, or a medical condition requiring radiation, chemotherapy or immunosuppression;
* Subjects who, in the opinion of the Investigator, would not be able or willing to comply with the protocol;
* Have a history of any autoimmune disease, such as, systemic lupus erythematosus (SLE), Addison's disease, Crohn's disease, multiple sclerosis or rheumatoid arthritis;
* Has had prior cervical spine surgery;
* Unstable cardiovascular, renal, hepatic, endocrine and/or pulmonary disease, cancer or uncontrolled diabetes;
* Have symptomatic disease requiring fusion of one level or > 2 levels and/or requiring fusion between levels C2-C4;
* Has cervical deformity secondary to acute or chronic traumatic fracture or neoplasm, including vertebral, facet or posterior element fracture or dislocation;
* Requires a concomitant posterior cervical surgery at the time of the ACDF;
* Has any contraindications for MRI;
* Is a ward of the state, prisoner, or transient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Swelling Index 1 Month | 1 month
  Difference of change from baseline to 1 month post operatively of soft tissue thickness/swelling, as measured by the swelling index on lateral x-rays.

SECONDARY OUTCOMES:
Swelling Index Other Timepoints | 3, 6 and 12 months
  Difference of change from baseline to discharge, 3, 6 and 12 months post operatively of soft tissue thickness/swelling, as measured by the swelling index on lateral x-rays
Neck Disability Index (NDI) Scores | 1, 3, 6 and 12 months
  The comparisons of score changes between groups at each timepoint will be investigated by employing linear regression
Visual Analog Scale (VAS) Scores | 1, 3, 6 and 12 months
  The comparisons of score changes between groups at each timepoint will be investigated by employing linear regression
Swallowing Quality of Life Questionnaire (SWAL-QOL) Scores | 1, 3, 6 and 12 months
  The comparisons of score changes between groups at each timepoint will be investigated by employing linear regression
Air Index Scores | 1, 3, 6 and 12 months
  The comparisons of score changes for 1, 3, 6, and 12 months from baseline will be investigated by using linear regression
Revision Surgery | 1, 3, 6 and 12 months
  The numbers and percentages of patients who underwent revision surgery as of each timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- Spine Institute of San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers